CLINICAL TRIAL: NCT00403871
Title: Anaesthetic Management of Women With Heart Disease For Labor and Delivery
Status: Completed | Type: Observational
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Other Study IDs: 06-05; 02-0211-E
Record Dates: First submitted 2006-11-23; First posted 2006-11-27 (Estimated); Last update posted 2007-03-02 (Estimated); Status verified 2007-02

CONDITIONS: Heart Diseases; Pregnancy
Keywords: Anaesthesia; Pregnency; Heart disease
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Heart disease among pregnant women is increasing in incidence. The cardiovascular changes associated with pregnancy may be particularly hazardous for both mother and fetus in a subset of these patients. The period of greatest risk is peripartum while these patients are under the care of the obstetrician and anesthesiologist. We will evaluate the anesthetic management of all women with heart disease whose pregnancies were followed at the University Health Network and/or Mount Sinai Hospital between 1986 and 2001.

DETAILED DESCRIPTION:
Heart disease among pregnant women is increasing in incidence. The cardiovascular changes associated with pregnancy may be particularly hazardous for both mother and fetus in a subset of these patients. The period of greatest risk is peripartum while these patients are under the care of the obstetrician and anesthesiologist. Exposing a compromised patient to general anesthesia is further complicated by the cardiovascular stress response to intubation and surgery, the cardiorespiratory implications of mechanical ventilation, the cardiac depression and vasodilation from general anesthetics, residual post-operative respiratory depression from general anesthetics and narcotics and the stress of weaning from mechanical ventilation and post-operative pain.

In the Adult Congenital Heart Program, obstetric patients are followed the by a specialized team of cardiologists, obstetricians and anesthesiologists who also follow all pregnant women referred with acquired cardiac disease. From this referral practice approximately 100 patients per year are now followed during their pregnancy and delivery. In conjunction with the ongoing system we intend to identify all parturients who delivered at the University Health Network (Toronto General Hospital) or Mount Sinai Hospital between the years 1986 and 2001. We will evaluate the anesthetic management of all women with heart disease whose pregnancies were followed at the University Health Network and/or Mount Sinai Hospital between 1986 and 2001.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with congenital or acquired heart disease
* Pregnant women with arrhythmias are also included providing they had had symptomatic tachyarrhythmias or bradyarrhythmias requiring treatment

Exclusion Criteria:

* Women with isolated mitral valve prolapse including those with mild to moderated mitral regurgitation
* Women referred for termination of pregnancy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 700
Dates: Start 2002-11; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Eric Goldszmidt, MD, Principal Investigator — Mount Sinai Hosiptal
Locations (2):
- Canada (2):
  - Mount Sinai Hospital, Toronto, Ontario
  - Univeristy Health Network, Toronto, Ontario